CLINICAL TRIAL: NCT00201019
Title: Improving Adherence to Blood Pressure Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 272; R01HL070740 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Active intervention participants receive a physician-pharmacist collaborative intervention.
  Interventions: Behavioral: Physician-pharmacist collaborative intervention
- 2 (No Intervention): Control participants do not receive recommendations from a clinical pharmacist.
- 3 (No Intervention): Passive intervention participants receive care by the same physicians caring for participants in the active intervention arm but are not seen by a clinical pharmacist. They are not actively enrolled in the study and do not have study visits for measuring blood pressure.

INTERVENTIONS:
Behavioral: Physician-pharmacist collaborative intervention — Participants receive assessment and medication and lifestyle recommendations from a clinical pharmacist.
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the impact of physician/pharmacist collaborative teams on hypertension guideline adherence for patients with uncontrolled hypertension in six family medicine practice sites in Iowa.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension is a prevalent chronic condition that, if left untreated, can lead to significant cardiovascular morbidity and premature mortality. There are established, evidence-based guidelines for the treatment of hypertension. However, these guidelines are not routinely adhered to by all providers for reasons that are not well known or understood. In addition, inadequate control of BP nationwide has been well documented. This study will explore barriers to guideline adherence (Phase I) and evaluate, via a randomized controlled trial, a new approach to enhancing guideline adherence and ultimately BP control.

DESIGN NARRATIVE:

The long-range goal of the principal investigator is to develop and evaluate collaborative relationships between physicians and pharmacists that improve pharmacotherapy. This will be a 5-year, multicenter study to evaluate the impact of physician/pharmacist collaborative teams on adherence to hypertension guidelines (JNC-VI) in six community-based family practice sites. There will be two study phases. Phase I comprises a needs assessment to identify barriers to guideline adherence and design intervention implementation refinement strategies. Phase II will be a prospective, randomized trial to assess the impact of physician/pharmacist collaborative teams on hypertension guideline adherence and BP control. The specific aims of Phase I are (1) to identify the scope and nature of physician and patient variables that may contribute to poor guideline adherence and (2) to refine the intervention implementation strategy and design tools for assessing guideline adherence and barriers to adherence. The specific aims of Phase II are (1) to determine if there is a change in guideline adherence and knowledge of hypertension when physicians are involved in physician/pharmacist teams and 2) to determine if physician/pharmacist teams can achieve better BP control compared to usual care. The investigators expect that the improvement in guideline adherence and reduction in BP with this intervention will significantly impact patients with hypertension. Because there are more than 37 million Americans with uncontrolled hypertension, this model has the potential to become an important strategy to help achieve the BP goals for Healthy People 2010.

ELIGIBILITY:
Inclusion Criteria for Phase II:

* Poorly controlled blood pressure based on clinic blood pressures
* Males or females, over 21 years of age
* Taking zero to three BP medications with no change in the regimen or dose within the past 4 weeks
* Have established medical care at the Family Medicine Clinic
* Nondiabetic patients with clinic BP values (average of the last three clinic readings during the previous 12 months) of 140 to 179 mm Hg systolic BP or 90 to 109 mm Hg diastolic BP, or diabetic patients with clinic BP values of 130 to 179 systolic or 80 to 109 diastolic

Exclusion Criteria for Phase II:

* Stage 3 hypertension (BPs greater than 180/110 mm Hg), or any evidence of hypertensive urgency or emergency
* Recent myocardial infarction or stroke (within the past 6 months prior to enrollment)
* New York Heart Association Class III or IV congestive heart failure
* Unstable angina
* Serious renal or hepatic disease, including greater than or equal to 1 gram of proteinuria per day
* Pregnancy
* Poor prognosis with a life expectancy estimated at less than 3 years
* Dementia or cognitive impairment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2003-08; Primary Completion 2008-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Adherence to hypertension guidelines | Measured for two 6 month periods: the first is prior to the participant's enrollment in the study and the second is while the participant is enrolled in the study

SECONDARY OUTCOMES:
Blood pressure control | Measured at baseline, 3 months, and 6 months
Physician knowledge | Measured prior to the start of the study and at the end of the study
Patient medication adherence | Measured at the time of enrollment and when the participant completes the study
Physician-pharmacist relationship | Measured prior to the start of the study and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Carter, PharmD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa College of Pharmacy, Iowa City, Iowa, United States

REFERENCES:
- [Background] Milchak JL, Carter BL, James PA, Ardery G. Measuring adherence to practice guidelines for the management of hypertension: an evaluation of the literature. Hypertension. 2004 Nov;44(5):602-8. doi: 10.1161/01.HYP.0000144100.29945.5e. Epub 2004 Sep 20. PMID 15381676
- [Background] Milchak JL, Carter BL, Ardery G, Black HR, Bakris GL, Jones DW, Kreiter CD. Development of explicit criteria to measure adherence to hypertension guidelines. J Hum Hypertens. 2006 Jun;20(6):426-33. doi: 10.1038/sj.jhh.1002005. PMID 16543909
- [Background] Carter BL, Hartz A, Bergus G, Dawson JD, Doucette WR, Stewart JJ, Xu Y. Relationship between physician knowledge of hypertension and blood pressure control. J Clin Hypertens (Greenwich). 2006 Jul;8(7):481-6. doi: 10.1111/j.1524-6175.2006.05601.x. PMID 16849901
- [Background] Carter BL. Antihypertensive prescribing: do we have reason to celebrate? Hypertension. 2006 Nov;48(5):816-7. doi: 10.1161/01.HYP.0000240978.77934.3a. Epub 2006 Sep 18. No abstract available. PMID 16982966
- [Background] Ardery G, Carter BL, Milchak JL, Bergus GR, Dawson JD, James PA, Franciscus C, Kim Y. Explicit and implicit evaluation of physician adherence to hypertension guidelines. J Clin Hypertens (Greenwich). 2007 Feb;9(2):113-9. doi: 10.1111/j.1524-6175.2007.06112.x. PMID 17268216
- [Background] Carter BL, Sica DA. Strategies to improve the cardiovascular risk profile of thiazide-type diuretics as used in the management of hypertension. Expert Opin Drug Saf. 2007 Sep;6(5):583-94. doi: 10.1517/14740338.6.5.583. PMID 17877445
- [Background] Carter BL, Rogers M, Daly J, Zheng S, James PA. The potency of team-based care interventions for hypertension: a meta-analysis. Arch Intern Med. 2009 Oct 26;169(19):1748-55. doi: 10.1001/archinternmed.2009.316. PMID 19858431
- [Derived] Carter BL, Ardery G, Dawson JD, James PA, Bergus GR, Doucette WR, Chrischilles EA, Franciscus CL, Xu Y. Physician and pharmacist collaboration to improve blood pressure control. Arch Intern Med. 2009 Nov 23;169(21):1996-2002. doi: 10.1001/archinternmed.2009.358. PMID 19933962